CLINICAL TRIAL: NCT05669495
Title: Remote Sleep Assessment in Adults at Risk for Dementia Using the ANNE Vital Sign System
Brief Title: ANNE Vital Sign System Remote Sleep Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Consortium on Neurodegeneration in Aging (Other)
Responsible Party: Sponsor
Other Study IDs: 5366
Record Dates: First submitted 2022-11-04; First posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment; Sleep Apnea
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No dementia, increased risk of dementia: Meets criteria for No Dementia and one of the following (according to CCNA Criteria):
  1. Cognitively Unimpaired
  2. Cognitively Unimpaired plus Subjective Cognitive Impairment
  3. Mild Cognitive Impairment (MCI)
  AND Classified as being at increased risk of dementia based on at least one of the following:
  1. First-degree family history of dementia
  2. Self-Reported or documented current and/or history at midlife (45-60 years) of the following risk factors:
  i. Hypertension ii. Hypercholesterolemia iii. Body Mass Index > 30 kg/m2 iv. Physical Inactivity v. Insomnia vi. Vascular-metabolic risk
  Interventions: Device: ANNE Vital Sign System

INTERVENTIONS:
Device: ANNE Vital Sign System — The ANNE Vital Sign System is a wireless remote monitoring system consisting of two flexible, soft, and skin-mounted electronic devices for use by researchers and healthcare professionals for continuous collection of physiological data in home and professional healthcare settings. The ANNE Vital Sign System integrates simultaneous synchronized ambulatory measurement of electrocardiography, photoplethysmography with derived pulse oximetry, pulse arrival time with derived beat-to-beat blood pressure, triaxial accelerometry, respiratory rate, and temperature, which would enable accurate measurement of sleep apnea. Indeed, in compelling in-laboratory preliminary data, we show the capacity for the ANNE Vital Sign System to detect and characterize sleep apnea in older patients. The ANNE Vital Sign System is non-invasive, flexible, easy to use, comfortable, and skin safe.

SUMMARY:
Sleep apnea is characterized by temporary pauses or stops to participant's breathing. Currently, sleep apnea is diagnosed using an in-lab sleep study, which involves spending a night in a sleep laboratory hooked up to wires on the head, chest, and legs. However, this is not feasible for many older adults. To overcome this barrier, the investigators will utilize an investigational vital signs monitor - the Advanced NeoNatal Epidermal (ANNE) Vital Sign System (Sibel Health, Evanston, IL,USA).

The primary objective of this study is to test the hypothesis that sleep apnea is associated with accelerated cognitive decline in older adults at risk for dementia. The investigators will measure sleep apnea at baseline and 12 months later and relate this to cognitive function at the same time points.

Sex-stratification will be used in analyses as appropriate. Qualitative feedback forms will be used to collect information about participant ease of use and experience with the ANNE Vital Sign System.

DETAILED DESCRIPTION:
Over 500,000 Canadians are currently living with dementia and this is predicted to reach one million in the next two decades. With no effective cures, there is an urgent need to identify and treat causal risk factors. Sleep and circadian rhythm disruption, including sleep deprivation, sleep fragmentation, sleep apnea, and abnormal circadian rhythms, are common. In model organisms, they accelerate development of dementia-associated neuropathologies and accumulating evidence suggests that in older adults they may be associated with a greater risk of dementia and dementia-related structural brain changes.

Sleep apnea is characterized by recurrent episodes of absent (apneas) or reduced (hypopneas) airflow in sleep, accompanied by hypercarbia and hypoxemia, and terminated by arousal and resumption of normal breathing. Sleep apnea is common in adults with Alzheimer's Disease (AD) and other dementias. The prevalence of moderate sleep apnea (apnea hypopnea index (AHI) > 15) in patients with mild AD is estimated at 68% and may be higher in moderate to severe AD. Moreover, a recent meta-analysis suggested that patients with AD have a five-fold increased odds of presenting with sleep apnea than adults with normal cognition.

The overall goal of this study is to test the hypothesis that sleep apnea is associated with accelerated cognitive decline in older adults at risk for dementia. The investigators will measure sleep apnea and its cardiovascular consequences at baseline and 12 months later and relate this to cognitive function at the same time points. To achieve this, the investigators will study participants enrolled in the Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia (CTU) and affiliated trials. The CTU is a Canada-wide study of older adults at risk for dementia, being undertaken by the Canadian Consortium on Neurodegeneration that will begin recruitment in May 2022. It, and affiliated trials, are anticipated to recruit 750 participants from May 2022-April 2024.

In clinical practice, sleep apnea is diagnosed using inpatient polysomnography. However, this is not feasible for many older adults. To overcome this barrier, the investigators will utilize an investigational vital signs monitor - the Advanced NeoNatal Epidermal (ANNE) Vital Sign System (Sibel Inc., Evanston, IL, USA).

The ANNE Vital Sign System is a wireless remote monitoring system consisting of two flexible, soft, and skin-mounted electronic devices for use by researchers and healthcare professionals for continuous collection of physiological data in home and professional healthcare settings. The ANNE Vital Sign System integrates simultaneous synchronized ambulatory measurement of electrocardiography, photoplethysmography with derived pulse oximetry, pulse arrival time with derived beat-to-beat blood pressure, triaxial accelerometry, respiratory rate, and temperature, which would enable accurate measurement of sleep apnea. Indeed, in compelling in-laboratory preliminary data, the investigators show the capacity for the ANNE Vital Sign System to detect and characterize sleep apnea in older patients. The ANNE Vital Sign System is non-invasive, flexible, easy to use, comfortable, and skin safe.

A separate 8-site Canadian in-lab study of the ANNE Vital Sign System is already underway, with participants undergoing diagnostic polysomnography per usual care or in the context of existing research projects approved by an institutional ethics board. ANNE Vital Sign System has an approved Investigational Testing Authorization (ITA) for this in-lab study (ITA application number 319430, approved December 11, 2020).

CTU recruiting sites will refer potential participants to Sunnybrook Research Institute (SRI) to obtain informed consent and then prepare shipment of ANNE Vital Sign System and instructions to participant. After study equipment and materials are shipped to and received by the participant, study staff will instruct the participant on the proper application and use of the ANNE Vital Sign System over remote video-conference. Specifically, study staff will instruct the participant to attach the two sensors of the ANNE Vital Sign System according to manufacturer recommendations. Participants will wear the sensors for 24 hours before removing it themselves at home and shipping back to Sunnybrook Research Institute. This procedure will be completed at two time points: Baseline and 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* The only inclusion criteria for this study is that participants must have consented and enrolled into a CTU affiliated study. There are no additional inclusion criteria. Individuals from CTU affiliated studies will be asked to confirm their enrollment in a CTU affiliated study as part of the informed consent process for this study.

For reference, inclusion criteria of CTU affiliated studies from which we will recruit may include, but are not limited to, the following list:

1. Ages 60-85
2. Sufficient proficiency in English or French
3. Technical ability to participate in remote assessments
4. Meets criteria for No Dementia and one of the following (according to CCNA Criteria):

   1. Cognitively Unimpaired
   2. Cognitively Unimpaired plus Subjective Cognitive Impairment
   3. Mild Cognitive Impairment (MCI)
5. AND Classified as being at increased risk of dementia based on at least one of the following: a. First-degree family history of dementia b. Self-Reported or documented current and/or history at midlife (45-60 years) of the following risk factors: i. Hypertension ii. Hypercholesterolemia iii. Body Mass Index > 30 kg/m2 iv. Physical Inactivity v. Insomnia vi. Vascular-metabolic risk

Exclusion Criteria:

1. Known nickel allergy
2. Known cardiac implantable device
3. Known arrhythmias
4. Otherwise unable to use the sensors; for example, finger amputations

For reference, exclusion criteria of CTU affiliated studies from which we will recruit may include, but are not limited to, the following list:

1. Participants who, in the opinion of the investigator, are not able to complete trial procedures remotely or adhere to the schedule of study assessments.
2. Individuals where English or French is not sufficiently proficient for remote clinical assessment.
3. Individuals who do not have the technical ability. Technical ability is defined as having computer and internet access; ability to send and receive emails; ability to participate in remote assessments.
4. Individuals who have a clinical diagnosis of Dementia
5. Clinical Dementia Rating (CDR; telephone/video-conference administration) Score of >1 or having a diagnosis of dementia based on DSM-IV criteria
6. Total Score on the Montreal Cognitive Assessment (MoCA; video-conference administration) <13

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrolled participants in the Canadian Therapeutic Platform Trial for Multidomain Interventions to Prevent Dementia (CTU) and affiliated trials. All participants will be individuals ages 60-85 classified as Not Dementia according to Canadian Consortium for Neurodegeneration in Aging (CCNA) criteria and classified as being at increased risk of dementia.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | Baseline
  Number of times per hour breathing slows or stops
Apnea Hypopnea Index | 12-months
  Number of times per hour breathing slows or stops
Oxygen Desaturation Index | Baseline
  Number of times per hour oxygen dips 4% or more
Oxygen Desaturation Index | 12-months
  Number of times per hour oxygen dips 4% or more
Hypoxemia Burden | Baseline
  integral area under the desaturation curve
Hypoxemia Burden | 12-months
  integral area under the desaturation curve
Time with oxygen saturation below 90% (O2<90) | Baseline
  As described in title
Time with oxygen saturation below 90% (O2<90) | 12-months
  As described in title

SECONDARY OUTCOMES:
Sex-stratification on Apnea Hypopnea Index | Baseline
  Sex-related effects on Apnea Hypopnea Index
Sex-stratification on Apnea Hypopnea Index | 12-months
  Sex-related effects on Apnea Hypopnea Index
Sex-stratification on Oxygen Desaturation Index | Baseline
  Sex-related effects on Oxygen Desaturation Index
Sex-stratification on Oxygen Desaturation Index | 12-months
  Sex-related effects on Oxygen Desaturation Index
Sex-stratification on Hypoxemia Burden | Baseline
  Sex-related effects on Hypoxemia Burden
Sex-stratification on Hypoxemia Burden | 12-months
  Sex-related effects on Hypoxemia Burden
Sex-stratification on Time with oxygen saturation below 90% (O2<90) | Baseline
  Sex-related effects on Time with oxygen saturation below 90% (O2<90)
Sex-stratification on Time with oxygen saturation below 90% (O2<90) | 12-months
  Sex-related effects on Time with oxygen saturation below 90% (O2<90)

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
LORIS is a web-based database solution for neuroimaging and other research data that is physically located at McGill University in Montreal. It will store data that has been processed to remove any direct identifiers of an individual study participant. Study subjects will be assigned a unique coded study identification number (LORIS Project Study Centre ID (PSCID)) that will be used to store their data. Local study sites will be responsible for storing all participant identifying information (name, contact, e-mail address) in secured encrypted databases and to maintain the master file that links the participant to their unique LORIS PSCID.
Supporting Information: Study Protocol, SAP
Time Frame: Duration of study

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT05669495/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT05669495/ICF_001.pdf